CLINICAL TRIAL: NCT06997055
Title: ROLL'YN-UST: Etude Observationnelle de Cohorte Pour la Prise en Charge Des Patients Atteints de Pathologies Inflammatoires Chroniques traités Par Steqeyma®, un Biosimilaire de l'ustékinumab
Brief Title: ROLL'YN-UST: an Observational Study in Patients Treated by Steqeyma®, an Ustekinumab Biosimilar
Acronym: ROLL'YN-UST
Status: Recruiting | Type: Observational
Sponsor: Celltrion HealthCare France (Industry)
Collaborators: Sanoia (Other)
Responsible Party: Sponsor
Other Study IDs: CTHC-CTP43-2; 2024-A02471-46 (Other: Ethics Committee Ouest I (Tours))
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Plaque Psoriasis
Keywords: Biosimilar; ustekinumab
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD group: Switch from ustekinumab originator in patients with Crohn's disease
  Interventions: Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg
- Psoriasis Group: Switch from ustekinumab originator in patients with Plaque Psoriasis
  Interventions: Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Ustekinumab 45 mg — biosimilar
Drug: Ustekinumab 90 mg — biosimilar

SUMMARY:
ROLL'YN-UST is a real-life study, which includes patients in clinical remission for at least 3 months and who have been treated with a reference biotherapy for at least 6 months, and for whom the physician has decided, independently of the study and as part of a shared medical decision, to switch them to STEQEYMA®. The main aim of this study is to the maintenance of clinical remission 12 months after initiation of a biosimilar as well as patient satisfaction 6 and 12 months after initiation of a biosimilar.

DETAILED DESCRIPTION:
Biotherapies have revolutionized the management of chronic inflammatory diseases in gastroenterology (Crohn's disease and ulcerative colitis), dermatology (e.g. plaque psoriasis and chronic spontaneous urticaria). However, due to their specificity and complexity, these treatments have a high financial cost, which has a significant impact on healthcare systems.

Following the loss of patent protection for these reference biotherapies, biosimilars were developed. These are similar to the reference molecules, but not strictly identical. As a result, to obtain marketing authorization, a biosimilar must demonstrate equivalence to the reference biologic in terms of efficacy and safety in a single indication defined in a Phase I (pharmacokinetic) and Phase III (clinical) study, before being extrapolated to other indications, as applicable.

This study aims to address these subjects for STEQEYMA® (CT-P43), a biosimilar ustekinumab approved by the European Commission on August 22, 2024, through a centralized procedure. STEQEYMA® is indicated for the treatment of moderate to severe forms of Crohn's disease (CD) and plaque psoriasis.

ROLL'YN-UST (CohoRt for the management Of chronic infLammatory diseases in a nationaL observational studY, in patieNts treated by Steqeyma®, an USTekinumab biosimilar - Etude observationnelle de cohorte pour la prise en charge des patients atteints de pathologies inflammatoires chroniques traités par Steqeyma®, un biosimilaire de l'ustekinumab) is a real-life study, which includes patients in clinical remission for at least 3 months and who have been treated with a reference biotherapy for at least 6 months, and for whom the physician has decided, independently of the study and as part of a shared medical decision, to switch them to STEQEYMA®. The main aim of this study is to the maintenance of clinical remission 12 months after initiation of a biosimilar as well as patient satisfaction 6 and 12 months after initiation of a biosimilar.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult (18 years of age or older at the time of inclusion) followed in specialty care and diagnosed with of one of the following conditions: Crohn's disease, Plaque psoriasis
* Treated for at least 6 months prior to inclusion with the reference Ustekinumab for the pathology in question: Crohn's disease, Plaque psoriasis
* Stable for at least 3 months according to the prescribing physician and in clinical remission according to the specific disease activity score.
* For whom the specialist has decided to switch to the biosimilar treatment developed and marketed by Celltrion on the day of inclusion (shared medical decision independent of the study)
* Have an email address.
* Have a mobile phone number.
* Be able to understand and complete questionnaires in French.
* Not opposed to participating in the study.
* Be affiliated to a French Social Security scheme or be a beneficiary of such a scheme.

Exclusion Criteria:

* Patients under guardianship or otherwise deprived of their freedom.
* Pregnant women or women of childbearing potential who wish to become pregnant while taking one of the study treatments.
* Patients participating at the time of inclusion in a clinical trial or other clinical study that prohibits simultaneous participation in other studies.
* Contraindication to study products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult dermatology or gastroenterology patients presenting a diagnosis for any of the following pathologies:
  * Crohn's Disease
  * Plaque Psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maintenance of remission, 12 months after initiation of biosimilar treatment | 12 months
  Percentage of patients still in clinical remission 12 months after initiation of biosimilar treatment according to the definitions used in the inclusion criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No